CLINICAL TRIAL: NCT05640934
Title: The Impact of Melatonin on the Postoperative Delirium in Geriatric Patients After Colorectal Surgeries. A Randomised Placebo-controlled Trial
Brief Title: Melatonin for Post Operative Delirium Prevention in Elderly Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Abd-Elazeem Abd-Elhameed Elbakry, Assistant professor, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 11/2022 ANEST10
Record Dates: First submitted 2022-11-29; First posted 2022-12-07 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Delirium in Old Age
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin group (Active Comparator): The patients will be given 5 mg melatonin the night before surgery, 12 hours before the scheduled time of surgery, followed by another 5 mg melatonin two hours before surgery.
  Interventions: Drug: Melatonin
- Control group (Placebo Comparator): The patients will be premedicated with placebo tablets, which will be administered at the same times as the melatonin group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin — The patients will be given 5 mg melatonin the night before surgery, 12 hours before the scheduled time of surgery, followed by another 5 mg melatonin two hours before surgery.
  Arms: Melatonin group
Drug: Placebo — The patients will be premedicated with placebo tablets, which will be administered at the same times as the melatonin group.
  Arms: Control group

SUMMARY:
The present study will evaluate the role of melatonin prophylaxis in delirium prevention in elderly patients undergoing colorectal procedures.

DETAILED DESCRIPTION:
This study is a prospective randomised double-blind placebo-controlled trial. Patients who meet the criteria for inclusion/exclusion will be evaluated. Melatonin tablets will be administered as a premedication to patients in the melatonin group. Patients in the control group will be given placebo tablets as a premedication. Fentanyl 1ug/kg and propofol 1-2 mg/kg will be used to induce anaesthesia. Atracurium 0.5 mg/kg will be used for the facilitation of endotracheal intubation. Isoflurane will be used to maintain anaesthesia and the depth of anaesthesia will be adjusted by a Bispectral index monitor. Postoperatively, the patients will be monitored for the development of delirium.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists (ASA) I to III physical status
* Elective colorectal procedures

Exclusion Criteria:

* Allergy to the research drugs,
* Patients who have vision or hearing impairment
* History of cerebral disorders
* Uncorrected acid-base, fluid, and electrolyte abnormalities
* History of central nervous system function affecting drugs.
* Chronic sedative-hypnotic administration at least one month prior to surgery
* Alcohol abuse
* Patients with recorded preoperative nursing delirium screening score ≥ 2.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-12-10 (Actual); Primary Completion 2023-07-02 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Incidence of delirium occurrence | Perioperative.
  Nursing delirium - screening score. It scores five items,Each item is rated from 0 to 2 where 0, absent; 1, mild; 2, severe. A score ≥ 2 is considered to have delirium.

SECONDARY OUTCOMES:
Degree of Sedation | Perioperative.
  Ramsay sedation score from 1 to 6. score 2 to 4 is acceptable sedation. Score 5 or 6 is excessive sedation
Intensity of pain | Perioperative
  Pain Assessment in Advanced Dementia Scale from 0 to 10 . score 1 to 3=mild pain; 4 to 6=moderate pain; 7-to 10=severe pain.
Mean arterial blood pressure | Perioperative
  mmHg
Heart rate | Perioperative
  beats/minute
Hypotension | Perioperative
  Number of patients with hypotension
Hypoxia | Perioperative
  Number of patients with hypoxia
Blood transfusion needs | Perioperative
  Number of patients needed blood transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Abd-Elazeem A Elbakry, MD, Principal Investigator — Menoufia University; Hazem E Elsersy, MD, Principal Investigator — Menoufia University; Islam M El-Desoky, MD, Principal Investigator — Menoufia University
Locations (1):
- Faculty of Medicine, Cairo, Shebin El-kom, Egypt

IPD SHARING:
Plan to Share IPD: No